CLINICAL TRIAL: NCT06716554
Title: Efficacy and Safety of Shatavari for Treatment of Menopausal Symptoms in Women: A Randomized, Double-blind, Three-arm, Parallel, Placebo-controlled Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SF Research Institute, Inc. (Network)
Collaborators: Ixoreal Biomed Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHT-1076-2024-1
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Menopause; Hot Flashes; Mood
MeSH Terms: conditions — Hot Flashes | interventions — Ashwagandha

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Shatavari (Experimental): One capsule of Shatavari 300 mg (contains Shatavari extract) once a day, orally with water.
  Interventions: Dietary Supplement: Shatavari extract
- Shatavari + Ashwagandha (Experimental): One capsule of Shatavari (300mg) + Ashwagandha (250mg) (contains Shatavari + Ashwagandha root extract) once a day, orally with water.
  Interventions: Dietary Supplement: Shatavari + Ashwagandha extract
- Placebo (Placebo Comparator): One capsule of Placebo 300 mg (contains starch extract) once a day, orally with water.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Shatavari extract — Shatavari is scientifically known as Asparagus racemosus. One capsule containing Shatavari 300mg should be taken once daily.
  Arms: Shatavari
Dietary Supplement: Shatavari + Ashwagandha extract — Shatavari is scientifically known as Asparagus racemosus along with Ashwagandha root extract scientifically known as Withania somnifera. One capsule containing Shatavari 300mg + Ashwagandha root extract 250mg should be taken once daily.
  Arms: Shatavari + Ashwagandha
Dietary Supplement: Placebo — Placebo (starch)
  Arms: Placebo

SUMMARY:
This is a Multi-center, Multi-national, Prospective, Randomized, Double-Blind, Placebo- Controlled three arm study to evaluate the efficacy and safety of Shatavari for the treatment of Menopausal symptoms in Women. Participants will be randomized to either one of the three treatment arms.Participants will then be asked to either take one capsule containing Shatavari or Shatavari + Ashwagandha or Placebo orally once daily in the morning after breakfast with a glass of water for 8 weeks. All the subjects will be asked to continue their routine diet and physical activities during the whole study period. The primary objective is to compare the efficacy of shatavari for treatment of menopausal symptoms in women. The secondary objective is to compare the safety of shatavari for treatment of menopausal symptoms in women.

DETAILED DESCRIPTION:
To qualify for the study, participants must be menopausal women aged 45 to 65 years with intact uterus and ovaries. Participants who complained of irregular menstrual cycle in the past 12 months, with a forward or postpone of a cycle more 7 days. At least 2 cycles were missing during the past 12 months, or reported menopause for at least 60 days. Women with complaints of menopausal symptoms, e.g., hot flash, insomnia, migraine, easy irritation, etc.

In this study, a maximum of 51 patients will be enrolled and the goal is to complete the study with at least 45 patients.

After signing this consent form, participants will answer questions regarding their medical history, including any medications they are taking. Physical exams with vital signs (pulse, temperature, sitting blood pressure and respiratory rate) will be performed at both visits by a professional trained to perform this testing.

It may be a Nurse (RN or LPN), Phlebotomist, or Medical Doctor. In order to be qualified to participate this study at initial Visit (Baseline), BMI score range between 18-35 are required.

A blood sample will be required from subjects. Subject's right or left arm will be used as the blood draw site, requiring a 5mL sample. The blood will be analyzing Sr. Estradiol, FSH, LH, Testosterone levels. These blood draws will be administered by a professional trained to perform this testing. It may be a Nurse (RN or LPN), Phlebotomist or Medical Doctor.

All eligible participants, will be given the required quantity of the study medication for self-administration, sufficient till the Visit 3- End of study visit, 8 weeks ± 4 Days. Participants will be randomized to either one of the three treatment arms.

Participants will be instructed to take one capsule of study medication to which they are randomized after breakfast, with ambient temperature water for 8 weeks at home. Participants will be asked to visit the site for Visit 2 (4 weeks ± 4 Days), Visit 3 (8 weeks ± 4 Days). Adverse events and concomitant medication will be recorded throughout the study. Participants will be asked to get used and unused study medications and their subject diaries in this visit. All the participants will be asked to continue their routine diet and physical activities during the whole study period.

The primary end point is the mean change in score for Menopause Rating Scale (MRS) from baseline. And the secondary end points are mean changes in scores for Perceived Stress Scale (PSS) questionnaire, Menopause Symptoms Treatment Questionnaire (MENQOL) scores, Profile of Mood States (POMS, abbreviated version) and mean changes in Serum hormones (Sr. Estradiol, FSH, LH, Testosterone) levels from baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Menopausal women aged 45 to 65 years with intact uterus and ovaries.
2. Participants who complained of irregular menstrual cycle in the past 12 months, with a forward or postpone of a cycle more 7 days. At least 2 cycles were missing during the past 12 months, or reported menopause for at least 60 days
3. Females with complaints of menopausal symptoms, e.g., hot flash, insomnia, migraine, easy irritation, etc.
4. Body mass index 18-35 kg/m2
5. Subject who has given written informed consent to participate in the study and understand the nature of the study
6. Able to read and write in English or any other vernacular language
7. No plan to commence new treatments over the study period.
8. Must have the ability and willingness to sign an informed consent and to comply with all study procedures.

Exclusion Criteria:

1. Participants taking any form of herbal extract in the last 3 months before study entry.
2. Participants who are on hormone replacement therapy (HRT) for more than 3 months.
3. Participants with Present active medical, surgical, and gynaecological problems.
4. Participants with a history of alcohol, tobacco dependence, or any substance abuse
5. Participants who had undergone bilateral ovariectomy
6. Participants with history of breast or cervical carcinoma
7. Participants who taking medication that affect bone metabolism, including glucocorticoid, anticonvulsant, and methotrexate.
8. Participants with Clinically relevant cardiovascular, gastrointestinal, hepatic, neurologic, endocrine, haematologic or other major systemic diseases making implementation of the protocol or other interpretation of the study result difficult
9. Participants with mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study
10. Participants with evidence of uncooperative attitude, including poor compliance.
11. Participants with inability to attend follow-up visit
12. Participants with any other medical condition (for example uncontrolled infection) that may, in the opinion of the Investigator, interfere with the study objective.
13. Patients with known hypersensitivity to Ashwagandha.
14. Patients who had participated in other clinical trials during the previous 3 months.
15. Patients who have any clinical condition, according to the investigator who does not allow safe fulfilment of clinical trial protocol

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Estimated)
Dates: Start 2024-10-26 (Actual); Primary Completion 2024-12-26 (Estimated); Study Completion 2025-01-20 (Estimated)

PRIMARY OUTCOMES:
Menopause Rating Scale (MRS) | MRS assessment will be done at Visit 1, Screening Visit/ Enrolment Visit/ Baseline Visit, (Day 1), Visit 2 (Week 4), and Visit 3- End of study visit, (Week 8).
  The scale consisted of 11 items, ranging from no symptoms to very severe symptoms. The total score of the MRS ranges from 0 (asymptomatic) to 44 (highest degree of complaints). The minimal/maximal scores vary between the three dimensions, depending on the number of complaints allocated to the respective dimension of symptoms.

SECONDARY OUTCOMES:
Perceived Stress Scale (PSS) | PSS assessment will be done at Visit 1, Screening Visit/ Enrolment Visit/ Baseline Visit, (Day 1), Visit 2 (Week 4), Visit 3 End of study visit, (Week 8).
  The Perceived Stress Scale (PSS-10) is the most widely used psychological instrument for measuring the perception of stress. It is a measure of the degree to which situations in one's life are appraised as stressful. Items were designed to tap how unpredictable, uncontrollable, and overloaded respondents find their lives. The scale also includes several direct queries about current levels of experienced stress. The questions in the PSS ask about feelings and thoughts during the last month. In each case, respondents are asked how often they felt a certain way
Menopause-Specific Quality of Life Questionnaire (MENQOL) | MENQOL assessment will be done at Visit 1, Screening Visit/ Enrolment Visit/ Baseline Visit, (Day 1), Visit 2 (Week 4), Visit 3 End of study visit, (Week 8).
  The MENQOL is self-administered and consists of a total of 29 items in a Likert-scale format. Each item assesses the impact of one of four domains of menopausal symptoms, as experienced over the last month: vasomotor (items 1-3), psychosocial (items 4-10), physical (items 11-26), and sexual (items 27-29). Items pertaining to a specific symptom are rated as present or not present, and if present, how bothersome on a zero (not bothersome) to six (extremely bothersome) scale.
Profile of Mood States (POMS, abbreviated version) | POMS assessment will be done at Visit 1, Screening Visit/ Enrolment Visit/ Baseline Visit, (Day 1), Visit 2 (Week 4), Visit 3 End of study visit, (Week 8).
  The POMS is a 40-item questionnaire rated on a 5-point Likert Scale, asking respondents how they feel right now. Scores are calculated for Tension, Anger, Fatigue, Depression, Esteem- related affect, Vigor, Confusion, and Total Mood Disturbance.
Serum Hormones | Blood samples for Serum hormones (Sr. Estradiol, FSH, LH, Testosterone) will be collected at Screening Visit/ Enrolment Visit/ Baseline Visit, (Day 1) and Visit 3- (Week 8)

CONTACTS AND LOCATIONS:
Locations (1):
- SF Research Institute, Inc., San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ademola J, Ajgaonkar A, Debnath T, Debnath K, Langade J. Efficacy and safety of Shatavari root extract (Asparagus racemosus) for menopausal symptoms: a randomized, double-blind, three-arm, placebo-controlled study. Front Reprod Health. 2025 Nov 27;7:1654503. doi: 10.3389/frph.2025.1654503. eCollection 2025. PMID 41394012